CLINICAL TRIAL: NCT00987220
Title: A Methodology Study To Evaluate Cerebrospinal Fluid Acetylcholine Following A Single Dose Administration Of Donepezil In Healthy Subjects
Brief Title: Effect of Aricept on Biomarkers (Acetylcholine, sAPP Alpha) In Cerebrospinal Fluid
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A9001428
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: CSF Biomarkers Acetylcholine
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, plasma, CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Placebo
  Interventions: Drug: Placebo
- donepezil (Aricept)
  Interventions: Drug: donepezil (Aricept)

INTERVENTIONS:
Drug: Placebo — Oral
  Groups: Placebo
Drug: donepezil (Aricept) — 5mg oral
  Other Names: Aricept
  Groups: donepezil (Aricept)

SUMMARY:
It is hypothesized that the acetylcholinesterase inhibitor, donepezil, will increase acute cerebrospinal fluid (CSF) actylcholine levels in healthy volunteers following a 5mg single dose oral administration.

DETAILED DESCRIPTION:
Sampling method based upon estimates of intra-subject biomarker variability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 18 to 33 kg/m2; and a total body weight >50 kg (110 lbs).
* Subject has the ability to understand the requirements of the study, provide written informed consent, and abide by the requirements of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of febrile illness within 5 days prior to the first study period.
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* A positive urine drug screen at screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first study period. As an exception, analgesics, caffeine, and non-pharmacological methods may be used on the discretion of the investigator to manage symptoms related to the lumbar catheterization. Aspirin, aspirin containing products, and non-steroidal anti-inflammatory agents that affect platelet function should not be used. Other exceptions may be granted by a qualified member of Pfizer study management.
* Treatment with an investigational drug within 30 days preceding the first study period.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception (as will be outlined in the protocol) from at least 14 days prior to enrollment in the study until completion of the study.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* Subjects with papilledema on exam at screening or on Day 0.
* Subject has any laboratory values outside the normal ranges on screening or on Day 0 which are deemed clinically significant by the investigator. Coagulation indices, including PT/aPTT, and platelet count must be normal.
* Subjects with lower spinal malformations, local infection, or other abnormalities that would exclude lumbar puncture (LP).
* Subjects who are unwilling or unable to comply with the Lifestyle guidelines presented in the protocol.
* Other severe acute or chronic medical or psychiatric condition/status or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results, and in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young (18-55) male and female healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Mean post-dose vs predose change in CSF acetycholine levels in donepezil compared to placebo control group. | 6 hrs

SECONDARY OUTCOMES:
Mean post-dose vs predose change in CSF histamine metabolites, sAPPalpha and inflammatory endpoints | 6hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001428&StudyName=Effect%20of%20Aricept%20on%20Biomarkers%20%28Acetylcholine%2C%20sAPP%20Alpha%29%20In%20Cerebrospinal%20Fluid%20